CLINICAL TRIAL: NCT03463642
Title: The Efficacy of Different Vitamin D Supplementation Delivery Methods on Serum 25(OH)D in Humans a Randomised Double-blind Placebo Trial
Brief Title: The Efficacy of Different Vitamin D Supplementation Delivery Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wolverhampton (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other); University of Worcester (Other)
Responsible Party: Principal Investigator, Matthew Wyon, Professor Matthew Wyon, University of Wolverhampton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UoW116976
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Mineral Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Vitamin D3 pill (Experimental): 100 pills = 100,000IU + Dicalcium phosphate, microcrystalline cellulose, silicium dioxide, magnesium stearate
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: Pill
- Pill placebo (Placebo Comparator): 100 pills = Dicalcium phosphate, microcrystalline cellulose, silicium dioxide, magnesium stearate
  Interventions: Dietary Supplement: Pill
- Vitamin D3 oral liquid (Experimental): 100 drops = 100,000IU in orange syrup
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: orange syrup
- Oral liquid placebo (Placebo Comparator): 100 drops orange syrup
  Interventions: Dietary Supplement: orange syrup
- Skin oil + Vitamin D3 + penetrator (Experimental): 100,000IU + mineral oil+ Tangerine essential oil (10ml)
  Interventions: Dietary Supplement: vitamin D3; Other: mineral oil; Dietary Supplement: Penetrator
- Skin oil + Vitamin D3 (Experimental): 100,000IU + mineral oil
  Interventions: Dietary Supplement: vitamin D3; Other: mineral oil
- Skin oil placebo (Placebo Comparator): Skin application: 100ml of mineral oil coloured with food colourant to match active oil sample
  Interventions: Other: mineral oil

INTERVENTIONS:
Dietary Supplement: vitamin D3 — 100,000IU
  Arms: Skin oil + Vitamin D3; Skin oil + Vitamin D3 + penetrator; Vitamin D3 oral liquid; Vitamin D3 pill
Dietary Supplement: Pill — Dicalcium phosphate, microcrystalline cellulose, silicium dioxide, magnesium stearate
  Arms: Pill placebo; Vitamin D3 pill
Dietary Supplement: orange syrup — 100 drops orange syrup
  Arms: Oral liquid placebo; Vitamin D3 oral liquid
Other: mineral oil — Paraffinum Liquidum,Isopropyl Palmitate,Parfum
  Arms: Skin oil + Vitamin D3; Skin oil + Vitamin D3 + penetrator; Skin oil placebo
Dietary Supplement: Penetrator — Tangerine essential oil (10ml)
  Arms: Skin oil + Vitamin D3 + penetrator

SUMMARY:
To test the efficacy of different vitamin D delivery methods on serum 25(OH)D. Participants randomly assigned to one of seven groups - three placebo groups and 4 active supplement groups receiving 100,000IU vitamin D3

DETAILED DESCRIPTION:
Various delivery methods of vitamin D supplementation are available to consumers but there have been no studies providing evidence of whether one delivery method is superior to others. The researchers wanted to compare the delivery of 100,000IU vitamin D3 by three methods on serum 25(OH)D levels. Two methods of oral supplementation (pill [prolonged release] and liquid [immediate release]), and delivery through the skin (with and without a penetrator enhancer. Placebo groups were pill, oral liquid and skin applied oil

ELIGIBILITY:
Inclusion Criteria:

* healthy, female

Exclusion Criteria:

* any participant that was taking vitamin supplementation, had a skin condition that would prevent them from applying oil to their skin or were taking, or had been taking in the past 6-months, oestrogen based contraception

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
serum 25(OH)D | 4 weeks
  Changes in serum 25(OH)D levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wolverhampton, Walsall, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Result] Stoll D, Dudler J, Lamy O, Hans D, Krieg MA, Aubry-Rozier B. Can one or two high doses of oral vitamin D3 correct insufficiency in a non-supplemented rheumatologic population? Osteoporos Int. 2013 Feb;24(2):495-500. doi: 10.1007/s00198-012-1962-5. Epub 2012 Mar 17. PMID 22426953
- [Result] Leventis P, Kiely PD. The tolerability and biochemical effects of high-dose bolus vitamin D2 and D3 supplementation in patients with vitamin D insufficiency. Scand J Rheumatol. 2009 Mar-Apr;38(2):149-53. doi: 10.1080/03009740802419081. PMID 18991184
- [Derived] Wyon MA, Wolman R, Martin C, Galloway S. The efficacy of different vitamin D supplementation delivery methods on serum 25(OH)D: A randomised double-blind placebo trial. Clin Nutr. 2021 Feb;40(2):388-393. doi: 10.1016/j.clnu.2020.05.040. Epub 2020 Jun 6. PMID 32703720